CLINICAL TRIAL: NCT04973761
Title: Evaliation of Oral Health Quality of Life for Children With Zirconium Crowns Versus Anteroir Strip Composite Crowns After 6 and 12 Months
Brief Title: Quality of Life for Children With Zirconium Anteroir Crowns Versus Strip Composite Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahmoud, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 401
Record Dates: First submitted 2021-07-17; First posted 2021-07-22 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strip composite crowns (Other)
  Interventions: Other: Strip composite crowns
- Zirconium crowns (Experimental)
  Interventions: Other: Zirconium crowns

INTERVENTIONS:
Other: Zirconium crowns — Prefabricated pirmary anteroir teeth zirconium crowns
  Arms: Zirconium crowns
Other: Strip composite crowns — Strip composite crowns
  Arms: Strip composite crowns

SUMMARY:
Early Childhood Oral Health Impact Scale (ECOHIS) will be used for detection of oral health related quality of life for children using strip composite crowns versus zirconium crowns at 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* healthy children Cariuos primary anteroir teeth Cooperative children

Exclusion Criteria:

* children with systemic diseases Children with bad oral habits

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Oral health related quality of life | 12 months
  Early Childhood Oral Health Impact Scale (ECOHIS).

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt